CLINICAL TRIAL: NCT04407273
Title: Statin Therapy and COVID-19 Infection (STACOV PROJECT)
Brief Title: Statin Therapy and COVID-19 Infection
Acronym: STACOV
Status: Completed | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Responsible Party: Principal Investigator, LUIS MASANA, MD, Dr, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: 106/2020
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: COVID; Statin; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with statins: Covid-19 infected patients with statins
  Interventions: Drug: observational
- without statins: Covid-19 infected patients without statins
  Interventions: Drug: observational

INTERVENTIONS:
Drug: observational — observational study

SUMMARY:
Considering that simvastatin, and probably statins in general, interfere with SARS-cov-2 cellular uptake and some inflammatory pathways activated by the virus, those patients on statin therapy should be less vulnerable to infection and their clinical course and prognosis should be better than that in individuals not on statin therapy.

DETAILED DESCRIPTION:
Statins reduce intracellular cholesterol synthesis by interfering with the limiting enzyme HMGCoA reductase. A lower intracellular cholesterol concentration leads to activation of the transcription factor SREBP 2 upregulating LDL receptor synthesis. In general, intracellular cholesterol homeostasis achieves a new physiological equilibrium at lower cholesterol concentrations. Moreover, the effect of cholesterol pathway inhibition has also an effect on farnesyl and geranyl molecules formation influencing protein prenylation leading to changes on inflammation and immunomodulation in vitro.

Changes in intracellular cholesterol alter cell membrane composition, particularly the structures referred to cholesterol rafts that accommodate a huge number of cell surface proteins as receptors. Theoretically, alterations in cholesterol rafts could derange the function of some receptors Some preliminary studies on cell models have suggested that statins could interfere the activity of some membrane viral receptors blunting its entry to cell (Berraondo P et al CIMA nonpublished data). SARS-cov-2 goes into cells through the Angiotensin Converser Enzyme 2 (ACE2) which is located in the surface of several cells including lung cells. It has been suggested that simvastatin could have a role in SARS-cov-2 infection by blocking the virus entry to cell. However, atorvastatin has been shown to increase ACE2 expression in animal models. Moreover, intracellular cholesterol content seems to influence the virus uptake.

Severe SARS-cov-2 infection is mediated by an inflammatory storm resulting in a deep tissue injury, endothelial damage, prothrombotic state and multiorgan failure. As mentioned above, statins also have some potent anti-inflammatory effects as modulating TNF, the NFkB transcription factor or blocking some members of the Tool Like Receptor family as TLR4-9 and its downstream cofactor MYD88. This anti-inflammatory effect has been implicated in a better prognosis of some diseases as HBV or HCV chronic infection, limiting the progression of hepatic damage to chronic liver disease or hepatocarcinoma. The impact of statin use on influenza epidemics has been repetitively assessed but contradictory or non-conclusive results have been obtained. The combination of statins and angiotensin receptor blockers have shown an important protective effect on other epidemics as Ebola, probably to their action on endothelium protection. A protective effect of statins on pulmonary hypertension development in a primate HIV model has also been reported. Although, in general all these pleiotropic effects of statins have been shown in vitro and its clinical impact is not clear, a clinical assay to test the efficacy of simvastatin on SARS-cov-2 is going on. Recently an observational study including more than 8000 patients infected by Sars-Cov-2 showed the protective effect of being on statins or ACE inhibitors. Taken into account its widespread use and putative effects on viral entry, inflammation, immune mechanisms and endothelial function, the use of standard therapies as statins have been postulated to target the host response to new virus pandemics.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old with a PCR or immunological confirmation of Covid-19 infection, admitted in the hospital for at least 24 hours, will be included.

Exclusion Criteria:

* Patients < 18 years old.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a retrospective observational multicentre study based on clinical records review.
  The following centres will take part in the study:
  LIPIDCAS Group:
  * Hospital Universitari Sant Joan
  * Hospital Universitari Joan XXIII
  * Hospital Sant Pau i Santa Tecla
  * Hospital Verge de la Cinta
  * Pius Hospital de Valls
  * Hospital del Vendrell
  Other centres from the LIPID AND ARTERIOSCLEROSIS UNITS NET (XULA) from Catalonia.
Sampling Method: Probability Sample
Enrollment: 2159 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
SARS-cov-2 scale of severity (9 steps) in Covid-19 infected patients with statin therapy | at the time of admission
  Assess the difference in the WHO SARS-cov-2 scale of severity (9 steps) achieved by Covid-19 infected patients, admitted in the hospital, with and without background statin therapy comparable in age and gender distribution

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Masana, Dr, Principal Investigator — Institut Investigacio Sanitaria Pere Virgili
Locations (1):
- Facultat de Medicina i Ciències de la Salut de Reus, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Masana L, Correig E, Rodriguez-Borjabad C, Anoro E, Arroyo JA, Jerico C, Pedragosa A, Miret M, Naf S, Pardo A, Perea V, Perez-Bernalte R, Plana N, Ramirez-Montesinos R, Royuela M, Soler C, Urquizu-Padilla M, Zamora A, Pedro-Botet J. Effect of statin therapy on SARS-CoV-2 infection-related mortality in hospitalized patients. Eur Heart J Cardiovasc Pharmacother. 2022 Feb 16;8(2):157-164. doi: 10.1093/ehjcvp/pvaa128. PMID 33135047

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/73/NCT04407273/Prot_SAP_000.pdf